CLINICAL TRIAL: NCT06652178
Title: Evaluation of Pelvic Floor Muscle Activity, Respiratory Functions, Respiratory Muscle Strength, and Functional Capacity in Children With Lower Urinary Tract Dysfunction
Brief Title: Pelvic Floor Muscle Activity, Respiratory Functions, Respiratory Muscle Strength, and Functional Capacity in Children With Lower Urinary Tract Dysfunction
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Deniz Tuncer, Assistant Professor, Bezmialem Vakif University
Other Study IDs: 31.05.2024-152562
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Lower Urinary Tract Disorder
Keywords: Lower Urinary Tract Disorder; Pelvic floor; Pulmonary Function; Respiratory muscle strength; Functional capacity; Children

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study Group: Children with lower urinary tract dysfunction
- Control Group: Healthy peers

SUMMARY:
The functional disorders of the lower urinary tract in children involve overactive bladder with thickening of the bladder muscle, resulting in a decrease in functional bladder volume and an increase in intra-bladder pressure. Lower urinary tract dysfunction in children most commonly develops due to non-neuropathic bladder sphincter dysfunction. Pelvic floor disorders is a term used to describe various diseases including mild, moderate and severe impairment of the pelvic floor muscles. Pelvic floor disorders become a condition that causes some symptoms such as involuntary urinary and faecal/gas incontinence, urgency and pelvic pain due to increased pressure of the pelvic floor muscles. Although the symptoms experienced may be permanent, they usually last throughout the day.

Electromyography (EMG) is a well-known non-invasive and practical method for relative pelvic floor muscle activity. Standardised endurance tests will be used for core muscle endurance measurements. Pulmonary function tests help to determine the severity of functional impairments and the extent to which treatment restores normal function. It has been reported that respiratory muscle strength tests can be used to monitor the effect of various diseases on muscle strength, especially considering their variations in the normal population. The six-minute walk test, which is used in the assessment of functional capacity, is frequently used in a wide range of different populations, including children, because it is easy to perform, has a low cost and especially shows exercise capacity. The six-minute walk test is an important indicator of aerobic endurance, which is one of the basic components of physical fitness.

The findings of this project will provide to see whether pelvic floor muscle activity, respiratory functions, respiratory muscle strength and functional capacity of children with lower urinary tract dysfunction differ from healthy children of the same age. The lack of a study on this subject suggests that this study would be an important contribution to the literature. In the present study, it was aimed to evaluate pelvic floor muscle activity with a superficial EMG device, core strength-endurance with core muscle endurance tests, respiratory functions with a spirometer (pulmonary function test), respiratory muscle strength (MIP/MEP) with an intraoral pressure measuring device, and functional capacity with a six-minute walk test. Determining how lower urinary tract dysfunction affects pelvic floor muscle activity, respiratory functions, respiratory muscle strength and functional capacity and the extent to which it affects the daily life of the individual is important. Furthermore, it is also considered that this project may provide valuable insight into how important it is to follow up the development of children with lower urinary tract dysfunction. The hypotheses of this study are as follows;

Hypotheses:

H1: Children with lower urinary tract dysfunction have poor pelvic floor muscle activity compared to healthy children.

H2: Children with lower urinary tract dysfunction have lower respiratory function than healthy children.

H3: Children with lower urinary tract dysfunction have lower respiratory muscle strength than healthy children.

H4: Children with lower urinary tract dysfunction have lower functional capacity than healthy children.

DETAILED DESCRIPTION:
Normal bladder function is essential for physical and psychosocial development in all children. The bladder has two main functions: storage and emptying. Bladder compliance is an important parameter for normal storage. For normal emptying, urinary continence until emptying and adequate emptying of stored urine under voluntary control are required. This task is achieved by coordination of the detrusor muscle of the bladder with the bladder neck or internal sphincter and voluntary external sphincter. Complete emptying of the bladder is achieved by adequate contraction. Incompatibility between the detrusor muscle and sphincter muscles may cause permanent damage by disrupting bladder functions. Lower urinary system dysfunction is categorized in three main groups as dysfunctional voiding, overactive bladder and underactive bladder. In addition, laughing incontinence, Hinman syndrome and vaginal reflux incontinence, which are rarely encountered, are also considered as lower urinary tract dysfunction. Lower urinary tract dysfunction in children is often due to non-neuropathic bladder sphincter dysfunction. Uninhibitable detrusor contractions (overactive bladder) and dysfunction of the pelvic floor muscles (dysfunctional voiding) are causes of lower urinary tract dysfunction. Lower urinary tract dysfunction is also defined as involuntary daytime urinary incontinence in children aged five years and older due to non-organic (functional) causes. Adequate bladder sphincter control and sphincter-detrusor compliance reach full maturity only around the age of four years. Normal daytime control of bladder function matures between 2-3 years of age, whereas nocturnal control is normally achieved between 3-7 years of age. It is known that symptoms of lower urinary tract dysfunction peak between 5-7 years of age. It has been shown in the literature that the frequency of lower urinary tract dysfunction is higher in patients with a family history. Especially if the mother or sibling has lower urinary tract dysfunction, the risk increases even more. Clinically, lower urinary tract dysfunction may present with various lower urinary tract symptoms such as urgency, urinary incontinence, frequent urination, dribbling and feeling of incomplete urinary emptying without an underlying uropathy or neuropathy. Studies have reported that the prevalence of lower urinary tract dysfunction is between 6-46%. Children with lower urinary tract dysfunction constitute 40% of the patients admitted to pediatric urology specialists. It is 5 times more common in girls than boys.

The pelvic floor muscles are divided into three layers consisting of deep, middle and superficial perineal muscles that extend from the symphysis pubis along the anterior lateral walls of the ilium towards the coccyx. The superficial layer includes bulbospongiosus, ischocavernosus, transversus perinei superfisialis and sphincter ani externus muscles; the middle layer includes sphincter urethra, external anal sphincter and transversus perinei profundus muscles. In the deep layer, there are levator ani and coccygeus muscles. The pelvic floor muscles are responsible for voiding, defecation, sexual function and support of the pelvic organs. In addition to these tasks, they also contribute to maintaining trunk stability. When the pelvic floor muscles contract, the perineum moves ventrally and cranially, closing the openings of the anus, vagina and urethra. These contractions are important in preventing involuntary leakage of urine and feces. A correct pelvic floor muscle contraction has been shown to increase urethral pressure. Pelvic floor dysfunction is an umbrella term characterized by different and complex symptoms.

Respiratory muscles and force ventilatory muscles are divided into two classes; primary and accessory muscles. The diaphragm is the main primary muscle and is active in normal breathing. The costae and diaphragm work together to produce three-dimensional changes in chest volume. During rest, only the inspiratory muscles are active. During exercise, the expiratory muscles also become active. The diaphragm contracts and flattens during normal respiration to allow inspiration; it then relaxes and returns to its resting shape during expiration. Vigorous expiration below the resting level also requires contraction of the abdominal muscles. The diaphragm, intercostal muscles, TA, multifidus and pelvic floor muscles are core stabilization muscles involved in postural function as well as being used for respiration. Daily physical activities require postural control and specific movement components. Many muscles in the core are important for postural smoothness and postural control during activities.

The diaphragm descends with inspiration to increase the pressure within the abdominal cavity, thus increasing the relaxation of the diaphragm, improving lung function and stabilizing the trunk. The pelvic floor muscle is activated by the increase in intra-abdominal pressure due to the action of the diaphragm, so that the TA muscle is easily activated by abdominal contraction during respiration. It shows that activation of the pelvic floor muscle and TA muscle facilitates stabilization of the thoracic cage and lumbar region and leads to improved respiratory function. These results suggest that it is important to ensure lumbar spine stabilization by increasing intra-abdominal pressure while focusing on diaphragmatic breathing and activation of core structures to transfer force from the center of the body to the lower extremities. It has been suggested that abdominal contraction during respiration activates the TA, external oblique, internal oblique and multifidus muscles more easily. Muscle tone of the diaphragm and TA muscle is particularly important to stabilize the lumbar region.

The diaphragm, TA and pelvic floor muscles are important for motor control, postural support and respiration. Their dysfunction results in back pain and an increased risk of injury. The respiratory function of these muscles needs to be integrated with many other functions such as swallowing, speech, valsalva maneuvers, spinal stabilization and trunk and limb movement. In situations of increased respiratory demand, such as stress, illness or physical exercise, the ability of the respiratory muscles to perform their postural tasks is reduced.

Spirometric measurement is the most widely used test of pulmonary function. It is a measurement of the maximum airflow to fill the lungs with sudden expiration after deep inspiration. It can provide information about the size of the airways (usually large airways) and the presence of obstructions in the airflow. The measurements obtained from spirometry are: FVC (forced vital capacity): The total volume of air that can be inhaled during a maximal forced expiration. FEV1: Forced expiratory volume in seconds is the volume expired in the first second of maximal expiration. FEV1/FVC: The ratio of volume expired in one second to FVC. PEF: Peak expiratory flow represents the maximum expiratory flow rate achieved. FEF25%-75%: The mean expired flow in the middle half of the FVC.

Respiratory muscle strength measurement methods are used to measure the strength of inspiratory and expiratory respiratory muscles. The most common areas of use are diagnosis, determination of severity and follow-up of respiratory muscle weakness. The easiest and most commonly used method to measure respiratory muscle strength is maximal inspiratory and expiratory intra-oral pressure measurements measured during airway opening with voluntary contraction against the closed airway. Maximal inspiratory intra-oral pressure (MIP) indicates inspiratory muscle force. After maximal expiration in the sitting position, the nose is closed with a nose clip and the person is asked to perform maximal inspiration for at least 1.5 s against the closed lid. The measurement is repeated 3 times and the highest value is taken. Maximal expiratory intraoral pressure (MEP) indicates expiratory muscle strength. After maximum inspiration in the sitting position, the person whose nose is closed with a nose clip is asked to perform maximum expiration for at least 1.5 s against the closed valve. The measurement is repeated 3 times and the highest value is taken.

The six-minute walk test, which is used in the assessment of functional capacity, is frequently used in a wide range of populations, including children, because it is easy to perform, low cost and especially because it also shows exercise capacity. The six-minute walk test is an important indicator of aerobic endurance, one of the main components of physical fitness.

The results the investigators will obtain with the project will allow to see how individuals with lower urinary tract dysfunction in children have an effect on pelvic floor muscle activity, respiratory functions, respiratory muscle strength and functional capacity compared to healthy individuals of the same age. Based on the lack of research on this subject and the lack of research on this subject in the literature, the study will make an important contribution to the literature. The investigators also think that this project can provide information on how important it is to follow the development of children with lower urinary tract dysfunction. The project is considered to fill an important gap in the literature in this regard. The aim with the project is to evaluate pelvic floor muscle activity, respiratory function, respiratory muscle strength and functional capacity in children with lower urinary tract dysfunction. In the study, it is aimed to measure pelvic floor muscle activity with a superficial EMG device, core strength-endurance with core muscle endurance tests, respiratory function with a spirometer (pulmonary function test), respiratory muscle strength (MIP/MEP) with an intraoral pressure measuring device, and functional capacity with a six-minute walk test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy lower urinary system without any dysfunction
* Being between the ages of 6-18
* Volunteering to participate in the study
* Not participating in a pelvic floor physiotherapy program for the last 6 months
* No intellectual and/or cognitive disability that would prevent participation in assessment and treatment

Exclusion Criteria:

* Having a disease related to the respiratory system
* Having a disease related to the musculoskeletal or neurological system
* History of abdominal, pelvic or spinal surgery

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The population of the study will consist of 14 volunteer subjects aged 6-18 years who are followed up by Bezmialem Vakıf University Faculty of Medicine, Department of Pediatric Urology with lower urinary tract dysfunction and 14 healthy controls in the same age group. All subjects will be evaluated and tested at Bezmialem Vakif University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Measurement of pelvic floor muscle activity | Day 1
  Electromyography (EMG) is a well-known noninvasive and practical method to measure pelvic floor muscle activity. Before the measurement, participants will be asked to urinate so that no urine remains in the bladder. The evaluator will position the participant in a supine position with the legs supported from underneath, knees flexed at 140 degrees, soles of the feet in contact with the bed, and thighs and feet approximately 30 centimeters apart. Participants will be taught to isolated contraction and relaxation of the pelvic floor muscles without using auxiliary muscles by palpation of the anus before EMG evaluation. Two superficial electrodes will then be placed bilaterally adjacent to the mucocutaneous line of the anus at the 2 and 7 o'clock positions. The reference electrode will be placed on the inner thigh. After proper placement of the electrodes, pelvic floor muscle activity will be measured. After rest, the participant will be asked to perform 5 consecutive seconds of maximal
Evaluation of pulmonary function-FVC% | Day 1
  Pulmonary Function Test will be performed with COSMED Pony FX (COSMED; Italy) spirometer in accordance with ATS/ERS criteria. Forced vital capacity (FVC) will be measured and expressed as percentage of predicted value.
Evaluation of pulmonary function-FEV1% | Day 1
  Pulmonary Function Test will be performed with COSMED Pony FX (COSMED; Italy) spirometer in accordance with ATS/ERS criteria. Forced expiratory volume in 1st second (FEV1) will be measured and expressed as percentage of predicted value.
Evaluation of pulmonary function-FEV1/FVC% | Day 1
  Pulmonary Function Test will be performed with COSMED Pony FX (COSMED; Italy) spirometer in accordance with ATS/ERS criteria. Forced Vital Capacity/Forced expiratory volume in 1st second (FEV1/FVC) will be measured and expressed as percentage of predicted value.
Evaluation of pulmonary function-PEF% | Day 1
  Pulmonary Function Test will be performed with COSMED Pony FX (COSMED; Italy) spirometer in accordance with ATS/ERS criteria. Peak Expiratory Flow (PEF) will be measured and expressed as percentage of predicted value.
Evaluation of pulmonary function- FEF25%-75% | Day 1
  Pulmonary Function Test will be performed with COSMED Pony FX (COSMED; Italy) spirometer in accordance with ATS/ERS criteria. The mean expired flow in the middle half of the FVC (FEF25%-75%) will be measured and expressed as percentage of predicted value.
Evaluation of respiratory muscle strength | Day 1
  Respiratory muscle strength will be measured with a portable, electronic intraoral pressure measuring device (MicroRPM, Micro Medical; UK) according to ATS/ERS criteria. Pressures will be assessed by measuring maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) during several seconds of maximal inspiration (Müller maneuver) and expiration (Valsalva maneuver) through the mouth.

SECONDARY OUTCOMES:
Evaluation of core muscle endurance-Trunk flexion test | Day 1
  The child's lower extremities will be placed as abducted at about shoulder-width, and the knees slightly flexed in supine position.
Evaluation of core muscle endurance-Trunk extension test | Day 1
  The child will be positioned in a prone position. The hips and ankles will be stabilized, the child will be asked to maintain the position, in which the trunk and legs are parallel to each other. The test will be terminated when the horizontal position can not be maintained (maximum 240 seconds).
Evaluation of core muscle endurance-Horizantal plank test | Day 1
  The child will be placed in the push-up position with shoulders and elbows in 90° flexion. The time keeping the body on their feet and forearms in a straight line will be recorded in seconds.
Evaluation of core muscle endurance-Side plank test | Day 1
  The child will be positioned in the side-lying position. The pelvis and trunk will be asked to be elevated to a horizontal position with support from the forearm and foot. Elevation will be performed on the forearm and ankle until the pelvis and trunk become horizontal. The time spent keeping the body in a straight line will be recorded in seconds.
Evaluation of functional capacity | Day 1
  Functional capacity will be assessed by the six-minute walk test according to ATS criteria. The distance covered by the participants in meters by walking as fast as possible at their own walking speed but without running for six minutes in a 30-meter straight corridor will be recorded in meters. In addition, SpO2, heart rate, dyspnea and fatigue levels will be evaluated by pulse oximetry (Beuer pulse oximeter, Beurer GmbH; Germany) before and after the test. Modified Borg Dyspnea and Fatigue Scales will be used to determine dyspnea and fatigue levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Istanbul, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Tuncer D, Arslanturk-Yildirim A, Yuvakgil EN, Ozturk H. Evaluation of pelvic floor muscle activity, pulmonary function, respiratory muscle strength, core muscle endurance, and functional capacity in children with lower urinary tract dysfunction. J Pediatr Urol. 2025 Dec;21(6):1543-1550. doi: 10.1016/j.jpurol.2025.08.027. Epub 2025 Aug 30. PMID 40935681